CLINICAL TRIAL: NCT06470477
Title: Molecular Characteristics of Phlegm-heat Syndrome in Ischemic Stroke: A Cohort Study
Brief Title: Molecular Characteristics of Phlegm-heat Syndrome in Ischemic Stroke
Status: Not yet recruiting | Type: Observational
Sponsor: Dongzhimen Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Ying Gao, Professor, Dongzhimen Hospital, Beijing
Other Study IDs: 82102823-02
Record Dates: First submitted 2022-11-14; First posted 2024-06-24 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Ischemic Stroke, Acute
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral blood will be collected at admission.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Phlegm-heat syndrome: Phlegm-heat syndrome: the score of "Phlegm-dampness syndrome" ≥10 and the score of "Internal fire syndrome" ≥10 in Diagnostic Scale for Syndrome Elements of Ischemic Stroke.
  Interventions: Drug: Guideline-based treatment
- Non-phlegm-heat syndrome: Non-phlegm-heat syndrome: the score of "Phlegm-dampness syndrome" <10 and the score of "Internal fire syndrome" <10 in Diagnostic Scale for Syndrome Elements of Ischemic Stroke.
  Interventions: Drug: Guideline-based treatment

INTERVENTIONS:
Drug: Guideline-based treatment — Guideline-based treatment includes anti-platelet therapy, control of vascular risk factors, and so on.
  Other Names: Routine care

SUMMARY:
The molecular characteristics of ischemic stroke with phlegm-heat syndrome and candidate biomarkers were identified based on multi-omics data. The main purpose of this study is to validate the molecular characteristics and biomarkers of phlegm-heat syndrome in ischemic stroke, and to demonstrate the association of biomarkers with clinical outcomes.

DETAILED DESCRIPTION:
This is a cohort study in patients with acute ischemic stroke. The demographic characteristics, Traditional Chinese Medicine (TCM) syndromes, and other baseline information will be recorded. At the same time, baseline peripheral blood will be collected. These participants will be followed up to 90 days of onset, and 90-day modified Rankin scale (mRS) scores will be assessed. The collected blood samples will be tested by multi-factor detection technology for candidate biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Acute ischemic stroke.
* Symptom onset within 72 hours.
* Diagnosis of phlegm-heat syndrome or non-phlegm-heat syndrome.
* Male or female ≥18 years and ≤ 80 years.
* With written informed consent.

Exclusion Criteria:

* Acute infectious diseases or acute exacerbations of chronic diseases within one month before enrollment.
* Patients has previous stroke.
* Other conditions that lead to motor dysfunction (e.g., severe osteoarthritis, rheumatoid arthritis).
* Renal or hepatic insufficiency, tumors, immune diseases, severe underlying diseases.
* Other conditions that affect the collection and evaluation of clinical information (e.g., severe aphasia, mental illness).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 to 80 years with acute ischemic stroke within 72 hours of onset.
Sampling Method: Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2024-06-20 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity, specificity, and area under the ROC curve of molecular features of Phlegm-heat syndrome in ischemic stroke | Baseline
  Sensitivity, specificity, and area under the ROC curve of molecular features of Phlegm-heat syndrome in ischemic stroke.
  The molecular characteristics of phlegm-heat syndrome in ischemic stroke include but are not limited to matrix metalloproteinase 9, mitogen-activated protein kinase 1, interleukin 6, and tumor necrosis factor.

SECONDARY OUTCOMES:
Proportion of patients independent | 90 days
  Proportion of patients independent is defined as the modified Rankin Scale score of 0, 1, or 2.
National Institute of Health Stroke Scale | Baseline, 7 days and 10 days after stroke onset.
  The National Institute of Health Stroke Scale (NIHSS) ranges from 0 to 42, with higher scores indicating more severe neurological deficits.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Gao, M.D., Principal Investigator — Dongzhimen Hospital, Beijing
Locations (1):
- Dongzhimen Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided